CLINICAL TRIAL: NCT04557449
Title: A PHASE 1/2A STUDY EVALUATING THE SAFETY, TOLERABILITY, PHARMACOKINETICS, PHARMACODYNAMICS, AND ANTI-TUMOR ACTIVITY OF PF-07220060 AS A SINGLE AGENT AND AS PART OF COMBINATION THERAPY IN PARTICIPANTS WITH ADVANCED SOLID TUMORS
Brief Title: Study to Test the Safety and Tolerability of PF-07220060 in Participants With Advance Solid Tumors
Acronym: CDK4i
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4391001; 2024-512120-11-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Liposarcoma; Prostate Cancer; Breast Neoplasms; Adenocarcinoma of Lung
Keywords: CDK4 inhibitor; Breast cancer; enzalutamide; fulvestrant; letrozole; endocrine therapy; Colorectal Cancer (CRC); Solid Tumors
MeSH Terms: conditions — Liposarcoma; Prostatic Neoplasms; Breast Neoplasms; Adenocarcinoma of Lung; Colorectal Neoplasms | interventions — Letrozole; Fulvestrant; Midazolam; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- 1A Monotherapy Escalation Arm 1 (Experimental): PF-07220060 Monotherapy Escalation
  Interventions: Drug: PF-07220060
- 1A Monotherapy Escalation Arm 2 (Experimental): PF-07220060 Monotherapy Escalation
  Interventions: Drug: PF-07220060
- 1A Monotherapy Escalation Arm 3 (Experimental): PF-07220060 Monotherapy Escalation
  Interventions: Drug: PF-07220060
- 1A Monotherapy Escalation Arm 4 (Experimental): PF-07220060 Monotherapy Escalation
  Interventions: Drug: PF-07220060
- 1B Combination Dose Finding Arm 1 (Experimental): PF-07220060 with Letrozole combination Escalation
  Interventions: Drug: PF-07220060; Combination Product: Letrozole
- 1B Combination Dose Finding Arm 2 (Experimental): PF-07220060 with Letrozole Combination Escalation
  Interventions: Drug: PF-07220060; Combination Product: Letrozole
- 1C Combination Dose Finding Arm 1 (Experimental): PF-07220060 with Fulvestrant Combination Escalation
  Interventions: Drug: PF-07220060; Combination Product: Fulvestrant
- 1C Combination Dose Finding Arm 2 (Experimental): PF-07220060 with Fulvestrant Combination Escalation
  Interventions: Drug: PF-07220060; Combination Product: Fulvestrant
- 2B Combination Dose Expansion (Experimental): PF-07220060 with Letrozole Combination Expansion
  Interventions: Drug: PF-07220060; Combination Product: Letrozole
- 2C Combination Dose Expansion (Experimental): PF-07220060 with fulvestrant Combination Expansion
  Interventions: Drug: PF-07220060; Combination Product: Fulvestrant
- 1D Monotherapy Food Effect (Experimental): PF-07220060 Monotherapy Food Effect
  Interventions: Drug: PF-07220060
- 1A Monotherapy Escalation Arm 5 (Experimental): PF-07220060 Monotherapy Escalation
  Interventions: Drug: PF-07220060
- 1F Combination Dose Finding (Experimental): PF-07220060 with Enzalutamide Escalation
  Interventions: Drug: PF-07220060; Combination Product: Enzalutamide
- 1E DDI Cohort (Experimental): PF-07220060 DDI with Midazolam
  Interventions: Drug: PF-07220060; Drug: Midazolam
- 2D Combination Dose Expansion (Experimental): PF-07220060 with enzalutamide Combination Expansion
  Interventions: Drug: PF-07220060; Combination Product: Enzalutamide
- 2A Combination Dose Expansion (Experimental): PF-07220060 with fulvestrant combination dose expansion
  Interventions: Drug: PF-07220060; Combination Product: Fulvestrant
- 2E Combination Dose Expansion (Experimental): PF-07220060 Monotherapy OR PF-07220060 plus fulvestrant combination therapy
  Interventions: Drug: PF-07220060; Combination Product: Fulvestrant

INTERVENTIONS:
Drug: PF-07220060 — CDK4 inhibitor
Combination Product: Letrozole — Endocrine Therapy
  Other Names: Femara
  Arms: 1B Combination Dose Finding Arm 1; 1B Combination Dose Finding Arm 2; 2B Combination Dose Expansion
Combination Product: Fulvestrant — Endocrine Therapy
  Other Names: Faslodex
  Arms: 1C Combination Dose Finding Arm 1; 1C Combination Dose Finding Arm 2; 2A Combination Dose Expansion; 2C Combination Dose Expansion; 2E Combination Dose Expansion
Drug: Midazolam — Benzodiazepine used for DDI
  Arms: 1E DDI Cohort
Combination Product: Enzalutamide — Androgen Receptor inhibitor
  Other Names: Xtandi
  Arms: 1F Combination Dose Finding; 2D Combination Dose Expansion

SUMMARY:
This is a Phase 1/2A, open label, multicenter, nonrandomized, multiple dose, safety, tolerability, pharmacokinetic and pharmacodynamic study of PF-07220060 administered as a single agent and then in combination with endocrine therapy.

The study consists of two parts and a China and Japan monotherapy cohort. Part 1 includes dose escalation cohorts evaluating PF-07220060 as single agent or in combination with endocrine therapy or enzalutamide, as well as a food effect cohort and a DDI cohort Part 2 includes dose expansion cohorts evaluating PF-07220060 in combination with endocrine therapy or enzalutamide.

In Part 1A, single escalating doses of PF-07220060 alone will be administered to determine the maximum tolerated dose (MTD) and select the recommended dose for expansion In Part 1B and Part 1C, PF-07220060 will be administered in combination with 1 of 2 endocrine therapies (letrozole and fulvestrant, respectively).

In Part 1D, food effect assessment of PF-07220060 at the RP2D dose level from the Part 1A will be conducted In Part 1E, the effect of PF-07220060 on the PK of midazolam will be evaluated (DDI) In Part 1F, escalating dosed of PF-07220060 will be administered in combination with enzalutamide Part 1B and Part 1C may commence at MTD or before reaching the MTD at a dose level in Part 1A.

Part 2A is a dose expansion cohort with fulvestrant and will explore more than one dose of PF-07220060 in participants diagnosed with mBC.

Part 2B and Part 2C are expansion for combination therapy of PF-07220060 with letrozole and fulvestrant, respectively.

Part 2D is the expansion cohort for combination therapy of PF-07220060 with enzalutamide.

Part 2E is an expansion cohort to evaluate PF-07220060 Monotherapy versus PF-07220060 plus fulvestrant combination therapy. The China monotherapy cohort will evaluate safety, tolerability and PK of PF-07220060 administered as single agent in Chinese participants.

The Japan monotherapy cohort will evaluate safety, tolerability and PK of PF-07220060 administered as a single agent in Japanese participants.

ELIGIBILITY:
Inclusion Criteria

* Part 1: Breast Cancer (BC)

  * Refractory Hormone Receptor Positive (HR+), Human Epidermal Growth Factor Receptor 2 Negative (HER2-) BC
  * Part 1A/Part 1D/Part1E also include: Refractory HR-positive/HER2-positive BC
* Part 1: Tumors other than BC (Part 1A/Part 1D/Part 1E): NSCLC, prostate, CRC, liposarcoma, or tumors with previously confirmed CDK4 or CCND1 amplification according to local standard tests
* Part 1F: prostate cancer
* Part 2A, 2B, 2C and 2E:

  * HR-positive/HER2-negative BC
  * Patients who are either postmenopausal women or pre/peri-menopausal (Part 2C only)
* Part 1D: metastatic castration resistant prostate cancer
* Lesion:

  * Part 1: evaluable lesion (including skin or bone lesion only)
  * Part 2A, 2B, 2C and 2E: measurable lesion per RECIST v1.1
  * Part 2D: Participants with evaluable disease as per PCWG3; participants with bone metastases only are allowed. Participants with biochemical recurrence only are excluded.
* Prior systemic Treatment

  * Part 1: HR-positive/HER2-negative BC

    * At least 1 line of SOC, including CD4/6 inhibitor therapy for advanced or metastatic disease, or if CDK4/6 inhibitors are not considered appropriate in the opinion of the investigator
    * At least 1 line of anti-endocrine in countries without CDK4/6 inhibitor approval or reimbursement, for advanced or metastatic disease
    * HR-positive/HER2-positive BC (Parts 1A/1D/1E): at least 1 prior treatment of approved HER2 targeting therapy
    * Tumors other than BC (Parts 1A/1D/1E/1F): tumor that is resistant to at least 2 lines of SOC for advanced or recurrent disease or for which no standard therapy is available
  * Part 2A and 2E: participants must have received at least 1 line of standard of care (including prior CDK4/6i) for advanced/metastatic disease; Prior chemo is allowed; Prior fulvestrant, mTOR and/or PI3K inhibitors are allowed
  * Part 2B: participants who have not received any prior systemic anti-cancer therapies for advanced/metastatic BC
  * Part 2C:

    * Progressed during treatment or within 12 months of completion of adjuvant therapy with an aromatase inhibitor if postmenopausal, or tamoxifen if pre or perimenopausal, or
    * Progressed while on or within 1 month after the endo the prior aromatase inhibitor therapy for advanced/metastatic BC if postmenopausal or prior endocrine treatment for advanced/metastatic BC if pre or perimenopausal
    * One previous line of chemotherapy for advanced/metastatic disease is allowed in addition to endocrine therapy
  * Part 2D:

    * Received prior abiraterone; enzalutamide and CDK4i naive
    * 0-1 line of chemotherapy is allowed General Inclusion Criteria
* All participants must be refractory to or intolerant of existing therapies known to provide clinical benefit for their condition.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* Adequate renal, liver, and bone marrow function

Exclusion Criteria:

* Part 1D: participants who have had a gastrectomy or have dietary or other restrictions that preclude a 10 hour overnight fast or consumption of the high fat, high calorie meal
* Part 2B: prior neoadjuvant or adjuvant treatment with a non-steroidal aromatase inhibitor with disease recurrence while on or within 12 months of completing treatment. Prior treatment with any CDK4/6 inhibitor
* Part 2C: prior treatment with any CDK inhibitor, fulvestrant, everolimus, or any agent whose mechanism of action is to inhibit the PI3K-mTOR pathway
* Known active uncontrolled or symptomatic Central Nervous System (CNS) metastases carcinomatous meningitis, or leptomeningeal disease
* Other active malignancy within 3 years prior to randomization, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ
* Major surgery or radiation within 4 weeks prior to study intervention
* Last anti-cancer treatment within 2 weeks prior to study intervention
* Participation in other studies involving investigational drug(s) within 4 weeks prior to study entry
* Pregnant or breastfeeding female participant
* Active inflammatory gastrointestinal (GI) disease, known diverticular disease or previous gastric resection or lap band surgery including impairment of gastrointestinal function or GI disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2026-09-23 (Estimated); Study Completion 2027-11-23 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities in the Dose Escalation Portion | Baseline up to day 28 of Cycle 1.
  First cycle (28 days) dose limiting toxicities (Parts 1A, 1B, 1C, 1F)
Incidence of clinically significant AEs | Weekly during Cycle 1 and 2 and then every 28 days through study completion, up to approximately 24 months; Each cycle is 28 days
  Adverse Events
Incidence of clinically significant laboratory assessments | Weekly during Cycle 1 and 2 (each cycle is 28 days) and then every 28 days through study completion, up to approximately 24 months
  safety laboratory abnormalities
Incidence of clinically significant abnormal vital and ECG parameters | Day 1, Day 8, Day 15 of Cycle 1 and starting from Cycle 2, and then every 28 days through study completion, up to approximately 24 months (Each cycle is 28 days)
  vital signs and heart rate corrected QT interval
Food Effect | Day -7 through the end of Cycle 1
  Maximal Concentration, Time to Maximum Plasma Concentration, Area under the Plasma Concentration (Part 1D)
DDI | D1 to the end of Cycle 1
  Maximal Concentration, Time to Maximum Plasma Concentration, Area under the Plasma Concentration (Part 1E)

SECONDARY OUTCOMES:
Single Dose: Maximal concentration (Cmax) in the Dose Escalation and Dose Finding portion | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Pharmacokinetic (PK) assessments for PF-07220060 (Parts 1A, 1B, 1C)
Single Dose: Time to Maximum Plasma Concentration (Tmax) in the Dose Escalation and Dose Finding portion | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Pharmacokinetic (PK) assessments for PF-07220060 (Parts 1A, 1B, 1C)
Single Dose: Area Under the Plasma Concentration Versus Time Curve from Time Zero to the Last Sampling Time Point Within the Dose Interval (AUClast) in the Dose Escalation and Dose Finding portion | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Pharmacokinetic (PK) assessments for PF-07220060 (Parts 1A, 1B, 1C)
Single Dose: Area Under the Plasma Concentration Versus Time Curve from Time Zero Extrapolated to Infinity (AUCinf) in the Dose Escalation and Dose Finding portion | Time Frame: Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Pharmacokinetic (PK) assessments for PF-07220060 (Parts 1A, 1B, 1C)
Apparent Oral Plasma Clearance (CL/F) in the Dose Escalation and Dose Finding portion | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Pharmacokinetic (PK) assessments for PF-07220060 (Parts 1A, 1B, 1C)
Single Dose: Apparent Volume of Distribution (Vz/F) in the Dose Escalation and Dose Finding portion | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Pharmacokinetic (PK) assessments for PF-07220060 (Parts 1A, 1B, 1C)
Multiple Dose: Steady State Maximal Concentration (Css,max) in the Dose Escalation and Dose Finding portion | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Pharmacokinetic (PK) assessments for PF-07220060 (Parts 1A, 1B, 1C)
Multiple Dose: Time to Maximum Plasma Concentration at Steady State (Tss,max) in the Dose Escalation and Dose Finding portion | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Pharmacokinetic (PK) assessments for PF-07220060 (Parts 1A, 1B, 1C)
Area Under the Plasma Concentration Versus Time Curve Within One Dose Interval (AUCss,t) in the Dose Escalation and Dose Finding portion | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Pharmacokinetic (PK) assessments for PF-07220060 (Parts 1A, 1B, 1C)
Multiple Dose: Steady State Minimum Plasma Concentration (Css,min) in the Dose Escalation and Dose Finding portion | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Pharmacokinetic (PK) assessments for PF-07220060 (Parts 1A, 1B, 1C)
Multiple Dose: Steady State Apparent Oral Plasma Clearance (CLss/F) in the Dose Escalation and Dose Finding portion | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Pharmacokinetic (PK) assessments for PF-07220060 (Parts 1A, 1B, 1C)
Multiple Dose: Apparent Volume of Distribution at Steady State (Vss/F) in the Dose Escalation and Dose Finding portion | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Pharmacokinetic (PK) assessments for PF-07220060 (Parts 1A, 1B, 1C)
Multiple Dose: Terminal Elimination Half-Life (t1/2) in the Dose Escalation and Dose Finding portion | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Pharmacokinetic (PK) assessments for PF-07220060 (Parts 1A, 1B, 1C)
Multiple Dose: Accumulation Ratio (Rac (AUCss,t /AUCsd,t)) in the Dose Escalation and Dose Finding portion | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Pharmacokinetic (PK) assessments for PF-07220060 (Parts 1A, 1B, 1C)
Tumor Response per RECIST v1.1 and per PCGW3 | baseline up to approximately 24 months
  Per RECIST v1.1 (Part 1 A-E; Part 2B and 2C); per PCWG3 (Part 1F and Part 2D)
Duration of Response (DOR) | baseline up to approximately 24 months
  Per RECIST v1.1
Progression Free Survival (PFS) | baseline up to approximately 24 months
  PFS per RECIST v.1.1
Time to Progression (TTP) | baseline up to approximately 24 months
  TTP per RECIST v1.1
Clinical Benefit Rate (CBR) | baseline up to approximately 24 months
  CBR per RECIST v1.1 (Parts 2B, 2C)
Peak and Trough Concentration of PF-07220060 | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Peak and trough concentration (Parts 2B, 2C, 2D)
Peak and trough concentrations of enzalutamide and N-desmethyl enzalutamide | Cycle 1 (each cycle is 28 days) and Day 1 of each subsequent cycle and at study completion visit, up to approximately 24 months
  Peak and trough concentrations (Part 2D)
Time to first skeletal events | Cycle 1 (each cycle is 28 days) to up to approximately 24 months
  Time to first skeletal events (Part 2D)
Quality of life questionnaire | Cycle 1 (each cycle is 28 days) to up to approximately 24 months
  time to functional status deterioration by FACT-P (Part 2D)
Radiographic Progression Free survival | Cycle 1 (each cycle is 28 days) up to approximately 24 months
  Part 2D
PSA50 | Cycle 1 (each cycle is 28 days) to up to approximately 24 months
  Part 1F and 2D

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- United States (11):
  - Ellison Institute, Los Angeles, California
  - Smilow Cancer Hospital at Yale - New Haven, New Haven, Connecticut
  - Yale-New Haven Hospital-Yale Cancer Center, New Haven, Connecticut
  - Smilow Cancer Hospital Phase 1 Unit, New Haven, Connecticut
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Institute- Chestnut Hill, Newton, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Sarah Cannon Research Institute - Pharmacy, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Argentina (5):
  - Hospital Británico de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Fundación Cenit Para La Investigación En Neurociencias, CABA, Ciudad Autã³noma de Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Clínica Universitaria Reina Fabiola, Córdoba
  - Fundación CORI para la Investigación y Prevención del Cáncer, La Rioja
- China (5):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Czechia (2):
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
- National Cancer Center Hospital East, Kashiwa, Chiba, Japan
- Mexico (6):
  - Hospital MAC Periferico Sur, Mexico City, Mexico City
  - INCAN, Mexico City, Mexico City
  - COI Centro Oncologico Internacional S.A.P.I. de C.V., Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Hospital Reforma, Oaxaca City, Oaxaca
  - Oaxaca Site Management Organization, Oaxaca City
- Slovakia (4):
  - Onkologicky ustav sv. Alzbety, s.r.o., Interna klinika VSZaSP a OUSA, Bratislava
  - Narodny onkologicky ustav, Bratislava
  - Fakultna nemocnica s poliklinikou Nove Zamky, Nové Zámky
  - POKO Poprad, s.r.o., Poprad
- United Kingdom (4):
  - Cancer Research UK Edinburgh Centre, Edinburgh, Edinburgh, CITY of
  - St Bartholomew's Hospital, London, London, CITY of
  - Sarah Cannon Research Institute UK, London
  - The Christie Hospital NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4391001